CLINICAL TRIAL: NCT02462057
Title: Testing the Effectiveness of Different Messaging Approaches to Increase Activation of a HealthyFood Benefit Amongst Individuals With Diabetes: A Randomised, Controlled Trial
Brief Title: Testing Different Messaging Approaches to Increase Activation of a HealthyFood Benefit in Adults With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Discovery Health (Industry)
Responsible Party: Principal Investigator, Anjali Gopalan, VA Advanced Fellow, Philadelphia VA Medical Center, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 821895
Record Dates: First submitted 2015-05-30; First posted 2015-06-03 (Estimated); Results first posted 2018-11-09 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-04

CONDITIONS: Diabetes; Diet; Incentives; Messaging
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Control Arm (No Intervention): This arm will represent current practice. This group will receive no contact from the research team. They may receive information regarding the benefit from the Vitality marketing team during the intervention period and can enroll in the benefit at any time during the study period.
- Diabetes-specific (Active Comparator): This group will receive a message which simply cites the two specific benefits of the eating more healthy foods for individuals with diabetes. This message contains a link to start the enrolment process.
  Interventions: Other: Email message regarding the HealthyFood benefit
- Experience of another member (Active Comparator): This group will receive a message that includes a quote from the perspective of a Vitality member with diabetes who uses the HealthyFood benefit. Given the need to standardise message content across study arms, the quote was written by the study team and not an actual member. The quote emphasizes the positive impact the benefit has had for the member-both the financial benefit, as well as the two specific diabetes health benefits.
  Interventions: Other: Email message regarding the HealthyFood benefit
- Input from a diabetes expert (Active Comparator): This group will receive a message that includes a quote from a South African physician who specializes in diabetes. The quote emphasises the financial benefit and the two specific diabetes health benefits of the HealthyFood program included in the other messages. It concludes with the doctor's recommendation of the benefit for all individuals with diabetes.
  Interventions: Other: Email message regarding the HealthyFood benefit
- Enhanced active choice (Active Comparator): This group will receive a message whose first portion is identical to those in the diabetes-specific message group. The second portion of the message differs in that instead of just asking recipients to click on the provided link if interested, the message asks people to choose and click on one of following possible responses:
  1. Yes! I want to active the HealthyFood benefit and get up to 25% cash back on the healthy food I buy at Pick n Pay or Woolworths
  2. No, I'd prefer not to activate and continue paying full price for my healthy food purchases
  Interventions: Other: Email message regarding the HealthyFood benefit

INTERVENTIONS:
Other: Email message regarding the HealthyFood benefit
  Arms: Diabetes-specific; Enhanced active choice; Experience of another member; Input from a diabetes expert

SUMMARY:
The Vitality HealthyFood benefit is a three-tiered incentive program designed to encourage healthier food choices amongst members of Discovery Health's Vitality program. Once enrolled in the benefit, participating members can receive 10%, 15%, or 25% cash-back on the healthy foods they purchase at selected grocers. And, while overall enrollment in the program is high, there is particular interest in increasing enrollment in the benefit amongst Vitality members with diabetes. One presumed barrier to enrollment in the benefit amongst members with diabetes is a misperception of the particular relevance of the benefit and healthier food choices for their personal health. Improved messaging regarding the HealthyFood benefit and its particular salience for individuals with diabetes may be an effective means of increasing activation of the benefit in this population. The proposed study will be a collaboration between Discovery Health/Vitality and researchers at the Perelman School of Medicine at the University of Pennsylvania. In the proposed RCT, Vitality members with diabetes will be randomised to different types of messages regarding the HealthyFood benefit. The investigators will then compare the effectiveness of these different messaging strategies at increasing activation of the HealthyFood benefit amongst Vitality members with diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over age 18
2. Vitality health members who have not yet enrolled in the Vitality HealthyFood benefit
3. Diagnosis of type 2 diabetes (based on registration for chronic benefits for type 2 diabetes)
4. Have registered on to Discovery Health/Vitality website in the past (marker of Internet access and availability of email address)

Exclusion Criteria:

* Anyone who does not meet above criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5467 (Actual)
Dates: Start 2015-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

REFERENCES:
- [Derived] Gopalan A, Paramanund J, Shaw PA, Patel D, Friedman J, Brophy C, Buttenheim AM, Troxel AB, Asch DA, Volpp KG. Randomised controlled trial of alternative messages to increase enrolment in a healthy food programme among individuals with diabetes. BMJ Open. 2016 Nov 30;6(11):e012009. doi: 10.1136/bmjopen-2016-012009. PMID 27903559

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5467 individuals were eligible in 1/2015. This sample was identified months before randomization to allow individuals time to learn about HF from other sources and enrol if interested. Prior to randomization, we excluded participants who joined HF of left Vitality since identification. This is why the initial and randomized samples are unequal.
Groups:
- Diabetes-specific: This group will receive a message which simply cites the two specific benefits of the eating more healthy foods for individuals with diabetes. This message contains a link to start the enrolment process.
  Email message regarding the HealthyFood benefit
- Experience of Another Member: This group will receive a message that includes a quote from the perspective of a Vitality member with diabetes who uses the HealthyFood benefit. Given the need to standardise message content across study arms, the quote was written by the study team and not an actual member. The quote emphasizes the positive impact the benefit has had for the member-both the financial benefit, as well as the two specific diabetes health benefits.
  Email message regarding the HealthyFood benefit
- Input From a Diabetes Expert: This group will receive a message that includes a quote from a South African physician who specializes in diabetes. The quote emphasises the financial benefit and the two specific diabetes health benefits of the HealthyFood program included in the other messages. It concludes with the doctor's recommendation of the benefit for all individuals with diabetes.
  Email message regarding the HealthyFood benefit
- Enhanced Active Choice: This group will receive a message whose first portion is identical to those in the diabetes-specific message group. The second portion of the message differs in that instead of just asking recipients to click on the provided link if interested, the message asks people to choose and click on one of following possible responses:
  1. Yes! I want to active the HealthyFood benefit and get up to 25% cash back on the healthy food I buy at Pick n Pay or Woolworths
  2. No, I'd prefer not to activate and continue paying full price for my healthy food purchases
  Email message regarding the HealthyFood benefit
Period: Overall Study
Arm/Group | Control Arm | Diabetes-specific | Experience of Another Member | Input From a Diabetes Expert | Enhanced Active Choice
Started | 791 | 793 | 812 | 752 | 758
Completed | 737 | 753 | 766 | 701 | 708
Not Completed | 54 | 40 | 46 | 51 | 50
Not completed — Left Vitality | 32 | 27 | 23 | 35 | 33
Not completed — Joined HealthyFood Before Intervention | 22 | 13 | 23 | 16 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Diabetes-specific | Experience of Another Member | Input From a Diabetes Expert | Enhanced Active Choice | Total
Number analyzed (Participants) | 737 | 753 | 766 | 701 | 708 | 3665
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (10.9) | 55.2 (10.7) | 55 (10.8) | 55.4 (10) | 56 (10.6) | 55.4 (10.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 145 | 152 | 152 | 134 | 146 | 729

OUTCOME MEASURES:

1. Primary Outcome: Enrollment in 10% Level of Benefit
Description: Rates of enrolment in 10% cash-back level (the most basic level, requires online activation only) of the HealthyFood Benefit amongst members with diabetes
Time Frame: One month from initial emailed messages
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Diabetes-specific | Experience of Another Member | Input From a Diabetes Expert | Enhanced Active Choice
Number analyzed (Participants) | 737 | 753 | 766 | 701 | 708
Participants | 7 | 57 | 76 | 48 | 89
Statistical Analysis 1: Comparison: Control Arm vs Diabetes-specific vs Experience of Another Member vs Input From a Diabetes Expert vs Enhanced Active Choice; Test type: Equivalence — The anticipated sample size of 3500 provided 80% power to detect a 3% pairwise difference between the proportions of participants who enrolled in HF with significance testing conducted at the Bonferroni-corrected significance level of 0.005 (0.05/10) to account for the 10 pairwise between-arm comparisons and pessimistically allowing for up to 10% further exclusions. The baseline monthly enrolment rate was estimated at ∼1%/month; p < 0.0001, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Control Arm | Diabetes-specific | Experience of Another Member | Input From a Diabetes Expert | Enhanced Active Choice
Serious Adverse Events (participants affected / at risk) | 0/737 | 0/753 | 0/766 | 0/701 | 0/708
Other Adverse Events (participants affected / at risk) | 0/737 | 0/753 | 0/766 | 0/701 | 0/708

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No